CLINICAL TRIAL: NCT06264414
Title: Phase III, Multicenter, Randomized, Double-blind Clinical Trial to Assess the Efficacy and Safety of the DTT106 in the Treatment of Erectile Dysfunction Associated With Benign Prostatic Hyperplasia
Brief Title: Efficacy and Safety of the DTT106 in the Treatment of Erectile Dysfunction Associated With Benign Prostatic Hyperplasia
Acronym: AUSTRÁLIA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTT106-III-0123
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Hyperplasia, Benign; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Hyperplasia; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DTT106 (Experimental): 1 hard capsule once a day, consistently 30 minutes after the same meal each day
  Interventions: Drug: DTT106
- dutasteride and tamsulosin (Active Comparator): 1 hard capsule once a day, consistently 30 minutes after the same meal each day
  Interventions: Drug: Dutasteride-Tamsulosin

INTERVENTIONS:
Drug: DTT106 — oral route
  Arms: DTT106
Drug: Dutasteride-Tamsulosin — oral route
  Arms: dutasteride and tamsulosin

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the DTT106 in the treatment of erectile dysfunction associated with benign prostatic hyperplasia

DETAILED DESCRIPTION:
After being informed about all risks and benefits and giving written informed consent, the subjects will undergo a 7-day screening to determine eligibility. After that, at visit 0 (V0), the subjects will be randomized to either the DTT106 or dutasteride + tamsulosin (0,5 mg + 0,4 mg).

ELIGIBILITY:
Inclusion Criteria:

* men aged 40 years and older.
* Sexually active men, with a defined partner, who have engaged in an average of 1 attempt at sexual intercourse per week in the last month.
* Participants under stable treatment with dutasteride + tamsulosin combination therapy.
* Diagnosis of erectile dysfunction, according to criteria established by the Guideline of the Brazilian Society of Urology and the American Society of Urology (2017);
* Erectile Function domain score of IIEF ≤ 25 and ≥ 6 points at the time of screening.

Exclusion Criteria:

* Any clinical or physical observation noted during evaluation by the investigating physician, or any laboratory condition, which is interpreted as posing a risk to participation in the clinical trial;
* Presence of uncontrolled chronic diseases;
* History of alcohol or illicit drug use disorder within the past 2 years;
* Men who are planning to impregnate their partners, or fertile men who are not using a reliable contraceptive method;
* Known allergy or hypersensitivity to the components of the medicinal products used during the clinical trial;
* History of pelvic surgery, prostatectomy, radiation therapy, penile implant placement surgery, urinary tract trauma, or invasive procedures for BPH treatment.
* Diagnosis of other diseases or conditions in the urinary tract, including, but not limited to: cancer, neurogenic bladder, urinary incontinence, recurrent infection, urethral stenosis, bacterial prostatitis.
* Clinical evidence of prostate cancer;
* Severe renal failure;
* Severe liver failure;
* Hypogonadism (supported by values below normal, as established by the local laboratory, for total testosterone) or absent libido (sex drive);
* Severe psychiatric or psychosocial disorders;
* Primary erectile dysfunction;
* Polyneuropathy, neurodegenerative diseases, spinal cord trauma or injury, tumors in the central nervous system, or other conditions that may affect erections;
* History of orthostatic hypotension.
* Expected to undergo cataract or glaucoma surgery;
* Concomitant use of any form of organic nitrate;
* Concomitant use of guanylate cyclase stimulators such as riociguat;
* Anatomical deformation of the penis that can significantly impair erection, including, but not limited to: angulation, cavernous fibrosis, and Peyronie's disease.
* Conditions that may predispose to priapism, including but not limited to: sickle cell anemia, multiple myeloma, leukemia;
* Prior diagnosis of pulmonary hypertension;
* Presence of anterior ischemic optic neuropathy, or degenerative diseases of the retina, including retinitis pigmentosa;
* Diagnosis of dysautonomia.
* Cardiovascular disease for which sexual activity is inadvisable, including but not limited to: Myocardial infarction in the last 90 days; Unstable angina or angina that occurs during sexual intercourse; Class 2 or higher heart failure according to the New York Heart Association in the last 6 months; Arrhythmias not controlled; Hypotension (< 90/50 mmHg) or uncontrolled hypertension; Stroke in the last six months.
* Diabetics with HbA1c greater than or equal to 10%, or with a history of retinopathy and/or neuropathy;
* Use of prohibited medications as per the protocol;
* Erectile dysfunction that has not responded to phosphodiesterase inhibitors type 5 (including but not limited to: sildenafil, tadalafil, vardenafil) at the time of screening.
* Participation in clinical trial protocols within the last 12 (twelve) months.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in the Erectile Function domain score of the International Index of Erectile Function (IIEF-EF) at the end of treatment, from baseline. | baseline and 12 weeks
  The IIEF (International Index of Erectile Function) is a quantitative measure used in the diagnostic assessment of erectile dysfunction. The IIEF is the sum of the scores assigned to each question, with scores ranging from 1 to 5, where 1=never and 5=always. The questionnaire covers five domains

SECONDARY OUTCOMES:
Change in maximum urinary flow rate (Qmax) | baseline and 12 weeks
  The maximum urinary flow rate (Qmax) will be measured by a flowmeter, compared to the baseline value, at the end of treatment
Decrease in post-void residual volume (PVR) | baseline and 12 weeks
  Change in post-void residual (PVR) volume, measured through prostate ultrasound
Improvement in urinary symptoms. | baseline and 12 weeks
  Change in the total International Prostate Symptom Score (IPSS) in patients.The IPSS relies upon the responses to seven questions regarding urinary symptoms and one question related to the patient's quality of life. Each question about urinary symptoms allows the patient to select one of six responses indicating the severity of the particular symptom. These responses are assigned points from 0 to 5. Consequently, the total score can vary from 0 to 35, with higher scores representing more severe symptoms. A higher score on the IPSS implies a poorer outcome.
Improvement in urinary emptying symptoms | baseline and 12 weeks
  Change in the score of the emptying domain of the IPSS (obstructive symptoms, questions 1, 3, 5, and 6). The IPSS relies upon the responses to seven questions regarding urinary symptoms and one question related to the patient's quality of life. Each question about urinary symptoms allows the patient to select one of six responses indicating the severity of the particular symptom. These responses are assigned points from 0 to 5. Consequently, the total score can vary from 0 to 35, with higher scores representing more severe symptoms. A higher score on the IPSS implies a poorer outcome.
Improvement in urinary storage symptoms. | baseline and 12 weeks
  Change in the score of the storage domain of the IPSS (irritative symptoms, questions 2, 4, and 7). The IPSS relies upon the responses to seven questions regarding urinary symptoms and one question related to the patient's quality of life. Each question about urinary symptoms allows the patient to select one of six responses indicating the severity of the particular symptom. These responses are assigned points from 0 to 5. Consequently, the total score can vary from 0 to 35, with higher scores representing more severe symptoms. A higher score on the IPSS implies a poorer outcome.
Improvement in the participant's quality of life in relation to their urinary condition | baseline and 12 weeks
  Change in the score of the quality-of-life item of the IPSS (IPSS-QoL). The IPSS relies upon the responses to seven questions regarding urinary symptoms and one question related to the patient's quality of life. Each question about urinary symptoms allows the patient to select one of six responses indicating the severity of the particular symptom. These responses are assigned points from 0 to 5. Consequently, the total score can vary from 0 to 35, with higher scores representing more severe symptoms. A higher score on the IPSS implies a poorer outcome.
Improvement in the participant's sexual function | baseline and 12 weeks
  Change in the total IIEF score. The 15-question IIEF Questionnaire is a validated, multi-dimensional, self-administered investigation found to be useful in the clinical assessment and treatment of erectile dysfunction. It examines the four main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. Each question is scored between 0 and 5, resulting in a total score range of 0-75 (higher score = less dysfunction). Higher scores indicate a better outcome.
Improvement in the participant's orgasmic function. | baseline and 12 weeks
  Change in the Orgasmic Function domain of the IIEF (IIEF-OF, questions 9 and 10). The 15-question IIEF Questionnaire is a validated, multi-dimensional, self-administered investigation found to be useful in the clinical assessment and treatment of erectile dysfunction. It examines the four main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. Each question is scored between 0 and 5, resulting in a total score range of 0-75 (higher score = less dysfunction). Higher scores indicate a better outcome.
Effectiveness of the treatment in improving the participant's sexual desire | baseline and 12 weeks
  Change in the Sexual Desire domain of the IIEF (IIEF-SD, questions 11 and 12). The 15-question IIEF Questionnaire is a validated, multi-dimensional, self-administered investigation found to be useful in the clinical assessment and treatment of erectile dysfunction. It examines the four main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. Each question is scored between 0 and 5, resulting in a total score range of 0-75 (higher score = less dysfunction). Higher scores indicate a better outcome.
Effectiveness in improving the participant's satisfaction with sexual relations | baseline and 12 weeks
  Change in the Satisfaction domain of Sexual Intercourse of the IIEF (IIEF-IS, questions 6, 7, and 8). The 15-question IIEF Questionnaire is a validated, multi-dimensional, self-administered investigation found to be useful in the clinical assessment and treatment of erectile dysfunction. It examines the four main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. Each question is scored between 0 and 5, resulting in a total score range of 0-75 (higher score = less dysfunction). Higher scores indicate a better outcome.
Overall satisfaction of the participant regarding their sex life. | baseline and 12 weeks
  Change in the General Satisfaction domain of the IIEF (IIEF-OS, questions 13 and 14). The 15-question IIEF Questionnaire is a validated, multi-dimensional, self-administered investigation found to be useful in the clinical assessment and treatment of erectile dysfunction. It examines the four main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. Each question is scored between 0 and 5, resulting in a total score range of 0-75 (higher score = less dysfunction). Higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- EMS, Hortolândia, São Paulo, Brazil